CLINICAL TRIAL: NCT02141594
Title: Diagnostic Ability of Posterior Pole Asymmetry Analysis Parameters (PPAA) of Spectralis Optical Coherence Tomography (OCT) in Detecting Early Glaucoma
Brief Title: Posterior Pole Asymmetry Analysis (PPAA) for Early Glaucoma
Acronym: PPAA
Status: Completed | Type: Observational
Sponsor: Dr T V Patel Eye Institute (Other)
Responsible Party: Principal Investigator, Paaraj Dave, Dr, Dr T V Patel Eye Institute
Other Study IDs: OCT PPAA in early glaucoma
Record Dates: First submitted 2014-05-14; First posted 2014-05-19 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Early glaucoma: The study group consisted of consecutive unilateral glaucoma patients, categorized as early stage by Hodapp-Anderson-Parrish classification.
- Normal subjects: Normal control subjects had a normal ocular examination, Intraocular pressure (IOP) <22 mmHg, no past history of high IOP, no family history of glaucoma, normal optic disc morphology and visual field in both eyes. One eye of control subject was randomly selected.

SUMMARY:
Spectrailis optical coherence tomography has come with a new posterior pole asymmetry analysis for glaucoma diagnosis. The aim of the investigators study was to assess its applicability in diagnosing early glaucoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 18 years
* Best corrected visual acuity 20/40 or better
* Refractive error within ±5D sphere and ±3D cylinder
* Willingness to participate in the study

Exclusion Criteria:

* Media opacities preventing imaging
* Intraocular surgery within the last 6 months
* Any retinal or neurological disease other than glaucoma that could confound the results of visual field examination and OCT.

Ages: 49 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive 80 eyes of 80 normal subjects and 76 eyes of 76 patients with early glaucoma were included for the study.
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2013-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Area under curve for all the diagnostic parameters of optical coherence tomography | up to 32 weeks
  This was a cross sectional study with one time measurement of the diagnostic parameters of the optical coherence tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Paaraj R Dave, MS, Principal Investigator — Dr TV Patel Eye Institute
Locations (1):
- Dr TV Patel Eye Institute, Vadodara, Gujarat, India

REFERENCES:
- [Result] Mori S, Hangai M, Sakamoto A, Yoshimura N. Spectral-domain optical coherence tomography measurement of macular volume for diagnosing glaucoma. J Glaucoma. 2010 Oct-Nov;19(8):528-34. doi: 10.1097/IJG.0b013e3181ca7acf. PMID 20164794
- [Result] Nakatani Y, Higashide T, Ohkubo S, Takeda H, Sugiyama K. Evaluation of macular thickness and peripapillary retinal nerve fiber layer thickness for detection of early glaucoma using spectral domain optical coherence tomography. J Glaucoma. 2011 Apr-May;20(4):252-9. doi: 10.1097/IJG.0b013e3181e079ed. PMID 20520570
- [Result] Seong M, Sung KR, Choi EH, Kang SY, Cho JW, Um TW, Kim YJ, Park SB, Hong HE, Kook MS. Macular and peripapillary retinal nerve fiber layer measurements by spectral domain optical coherence tomography in normal-tension glaucoma. Invest Ophthalmol Vis Sci. 2010 Mar;51(3):1446-52. doi: 10.1167/iovs.09-4258. Epub 2009 Oct 15. PMID 19834029
- [Result] Rao HL, Babu JG, Addepalli UK, Senthil S, Garudadri CS. Retinal nerve fiber layer and macular inner retina measurements by spectral domain optical coherence tomograph in Indian eyes with early glaucoma. Eye (Lond). 2012 Jan;26(1):133-9. doi: 10.1038/eye.2011.277. Epub 2011 Nov 11. PMID 22079964